CLINICAL TRIAL: NCT06140524
Title: Phase 2 Dose-Ranging and Interception Study of Linvoseltamab in Patients With High-Risk Monoclonal Gammopathy of Undetermined Significance or Non-High-Risk Smoldering Multiple Myeloma
Brief Title: A Proof-of-Concept Study to Learn Whether Linvoseltamab Can Eliminate Abnormal Plasma Cells That May Lead to Multiple Myeloma in Adult Patients With High-Risk Monoclonal Gammopathy of Undetermined Significance or Non-High-Risk Smoldering Multiple Myeloma
Acronym: LINKER-MGUS1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R5458-ONC-2257; 2023-505242-25-00 (EU CTIS Number)
Record Dates: First submitted 2023-10-31; First posted 2023-11-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-08

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance (MGUS); Smoldering Multiple Myeloma (SMM)
Keywords: linvoseltamab; monoclonal immunoglobulin (M-protein); cancer interception; immunotherapy; plasma cell disorders
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Safety Run-In (Part 1) (Experimental): Sequential groups of participants will be enrolled to assess the initial safety and tolerability of the step-up regimen leading up to the start of different full doses of linvoseltamab.
  Interventions: Drug: Linvoseltamab
- Expansion (Part 2) - Dose regimen 1 (Experimental): Participants will be randomized in a 1:1:1:1 ratio across 4 dosing regimens
  Interventions: Drug: Linvoseltamab
- Expansion (Part 2) - Dose regimen 2 (Experimental): Participants will be randomized in a 1:1:1:1 ratio across 4 dosing regimens
  Interventions: Drug: Linvoseltamab
- Expansion (Part 2) - Dose regimen 3 (Experimental): Participants will be randomized in a 1:1:1:1 ratio across 4 dosing regimens
  Interventions: Drug: Linvoseltamab
- Expansion (Part 2) - Dose regimen 4 (Experimental): Participants will be randomized in a 1:1:1:1 ratio across 4 dosing regimens
  Interventions: Drug: Linvoseltamab

INTERVENTIONS:
Drug: Linvoseltamab — Administered per the protocol
  Other Names: REGN5458; Lynozyfic™

SUMMARY:
This study is researching an investigational drug called linvoseltamab ("study drug") in participants at moderate risk of developing multiple myeloma (about 3 to 10% average annual risk), a group that consists of patients with precancerous conditions called High-Risk Monoclonal Gammopathy of Undetermined Significance (HR-MGUS) and Non-High-Risk Smoldering Multiple Myeloma (NHR-SMM).

The primary purpose of the study is to understand how well the study drug can eliminate abnormal plasma cells and laboratory signs of HR-MGUS and NHR-SMM.

The study is looking at several other research questions, including:

* How many participants treated with linvoseltamab have improvement of their HR-MGUS or NHR-SMM?
* What side effects may happen from taking the study drug?
* How much study drug is in the blood at different times?
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects).

ELIGIBILITY:
Key Inclusion Criteria:

1. HR-MGUS or NHR-SMM as defined in the protocol
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
3. Adequate hematologic and hepatic function, as described in the protocol
4. Estimated glomerular filtration rate (GFR) ≥30 mL/min/1.73 m^2 by the Modification of Diet in Renal Disease (MDRD) equation

Key Exclusion Criteria:

1. High-risk SMM, as defined in the protocol
2. Evidence of any of myeloma-defining events, as described in the protocol
3. Diagnosis of systemic light-chain amyloidosis, Waldenström macroglobulinemia (lymphoplasmacytic lymphoma), solitary plasmacytoma, or symptomatic MM
4. Clinically significant cardiac or vascular disease within 3 months of study enrollment, as described in the protocol
5. Any infection requiring hospitalization or treatment with intravenous (IV) anti-infectives within 28 days of the first dose of linvoseltamab
6. Uncontrolled Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection; or other uncontrolled infection or unexplained signs of infection, as described in the protocol

NOTE: Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2032-05-18 (Estimated); Study Completion 2032-05-18 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events Interest (AEI) during the safety observation period | 35 days
  Part 1 An AEI is a toxicity potentially related to study treatment that may preclude dose escalation or expansion according to the Bayesian Optimal Interval (BOIN) design decision rules
Frequency of Treatment-Emergent Adverse Event (TEAEs) during the safety observation period | 35 days
  Part 1 As assessed by the NCI-CTCAE grading system version 5 (for all grades)
Severity of TEAEs during the safety observation period | 35 days
  Part 1 As assessed by the NCI-CTCAE grading system version 5 (for all grades)
Achievement of Complete Response (CR) as determined by the investigator | Up to 5.5 years
  Part 2

SECONDARY OUTCOMES:
Frequency of TEAEs | Up to 5.5 years
  As assessed by the NCI-CTCAE grading system version 5 (for all grades)
Severity of TEAEs | Up to 5.5 years
  As assessed by the NCI-CTCAE grading system version 5 (for all grades)
Frequency of Serious Adverse Events (SAEs) | Up to 5.5 years
Severity of SAEs | Up to 5.5 years
Frequency of laboratory abnormalities | Up to 5.5 years
  As assessed by the NCI-CTCAE grading system version 5 (for all grades)
Severity of laboratory abnormalities | Up to 5.5 years
  As assessed by the NCI-CTCAE grading system version 5 (for all grades)
Minimal Residual Disease (MRD) negativity among participants that achieve a response of CR | Up to 5.5 years
Sustained MRD negativity on an annual basis | Up to 3 years after achievement of CR
Overall response of Partial Response (PR) or better as determined by the investigator | Up to 5.5 years
Duration Of Response (DOR) as determined by the investigator | Up to 5.5 years
Biochemical Progression-Free Survival (PFS) as determined by the investigator | Up to 5.5 years
Concentration of linvoseltamab in serum over time | Up to 9 months
Incidence of Anti-Drug Antibodies (ADAs) to linvoseltamab over the study duration | Up to 5.5. years
Magnitude of ADAs to linvoseltamab over the study duration | Up to 5.5. years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (13):
- United States (6):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health, Ann Arbor, Michigan
  - Stony Brook University Hospital, Stony Brook, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington
- Spain (7):
  - Hospital Universitario Virgen de las Nieves, Granada, Andalusia
  - Hospital Universitari Mutua Terrassa, Terrassa, Barcelona
  - Hospital Clinico Universitario Virgen De La Arrixaca, El Palmar, Murcia
  - Hospital de Cabuenes, Gijón, Principality of Asturias
  - Hospital Sant Pau, Barcelona
  - Universitaru Hospital La Princesa, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/